CLINICAL TRIAL: NCT03467269
Title: BRUSH Sign: Radiolographic Marker of Cerebral Infarctus Prognosis
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: BRUSH SIGN
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Brush sign — presence of a brush sign in MRI image in acute cerebral ischaemia

SUMMARY:
Today the treatment of ischemic stroke in acute phase is based on medicinal or endovascular revascularization. Cerebral MRI sequences help the diagnostic. This procedure uses deoxyhemoglobin as an endogenous tracer. This is also a scorer of cerebral ischemia and the increase lets visualized transcerebral veins in the suffering zone giving a brush aspect. Several studies show the interest of this sign and conclude that deoxyhemoglobin presence is a predictive factor of cerebral ischemia. The aim of the study is to evaluate this brush-sign and correlate it with the prognosis retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years old
* hospitalized for cerebral infarction
* MCA territory
* MRI within 24hours
* Sequence of magnetic susceptibility (SWAN)

Exclusion Criteria:

* Incomplete cerebral infarct
* MRI not possible

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient hospitalized between april 2014 and august 2016 for cerebral infarction
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
autonomy level | Month 3
  measurement of autonomy level by mRS

CONTACTS AND LOCATIONS:
Overall Officials: ZUBER Mathieu, Professor, Principal Investigator — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France